CLINICAL TRIAL: NCT04800835
Title: A Study to Compare the Safety and Effectiveness of the 12-month Spatz3 Adjustable Balloon With a 6-Month Non Adjustable Balloon in the Weight Management of Subjects
Brief Title: A Study to Compare the 12-month Spatz3 Adjustable Balloon With a 6-month Non Adjustable Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spatz FGIA, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sp12Or6
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Gastric Balloon

STUDY DESIGN:
Intervention Model Description: Subjects will be studied in a randomized open label single center study that will run 52 weeks. Subjects will be randomized to two treatment groups: Group 1- Spatz3 adjustable balloon 12-month implantation; and Group 2 - 6-month non adjustable balloon implantation with additional 6 months of dietician follow-up after balloon extraction
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Spatz3 adjustable balloon 12-month implantation; (Active Comparator): A 12 month adjustable intragastric balloon for weight loss that can have the balloon volume increased or decrease as needed
  Interventions: Device: Gastric Balloon
- Group 2- 6-month non adjustable balloon implantation with additional 6 months follow-up (Active Comparator): A 6-month non adjustable intragastric balloon for weight loss
  Interventions: Device: Gastric Balloon

INTERVENTIONS:
Device: Gastric Balloon — implantation of two types of gastric balloons. Spatz3 Adjustable balloon will be implanted for 12 months and 6-month non adjustable balloon will be implanted for 6 months

SUMMARY:
The purpose of this study is to compare a 12-month adjustable balloon over a 6-month non-adjustable balloon with 6-month dietician follow-up. The endpoint is %TBL at 12 months.

DETAILED DESCRIPTION:
Subjects will be studied in a randomized open label single center study that will run 52 weeks. Subjects will be randomized to two treatment groups: Group 1- Spatz3 adjustable balloon 12-month implantation; and Group 2 - non adjustable 6-month implantation with additional 6 months of dietician follow-up after balloon extraction. Fourth four eligible subjects will be randomized to treatment groups 1 and 2 and will undergo endoscopy and implantation of either the Spatz3 Adjustable Balloon or the 6-month non adjustable Balloon. All subjects will follow a calorie restricted diet designed by the dietician. The initial diet will be liquid and will be advanced as per the dietician's recommendations. Changes in diet will depend on subject tolerance to the balloon and specific food intolerances and will be adjusted frequently by the dietician. The initial balloon volume will be 500 ml of 0.9% normal saline with 2 ml of a 1% solution of methylene blue. An adjustment will be performed for treatment Group 1 at Week 24 (±6 weeks) with the addition of 200-300 ml of 0.9% normal saline, as per section 1.6.2.1.3.3. The balloon adjustment procedure is done with an endoscopy procedure under the same sedation as the implantation procedure. The subjects will have follow up by the PI/Nurse Practitioner and the Dietician/Nutritionist periodically as per section 1.7.3. until extraction at 52 weeks. The 6-month non adjustable balloon treatment group will undergo balloon extraction at 6 months followed by monthly dietician vists for an additional 6 months. The study will terminate at the end of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have a BMI ≥ 27
2. Be male or female, between 18 and 65 years of age, inclusive;
3. Have a history of excess weight (BMI ≥ 27 kg/m2) for at least 2 years and have failed more conservative weight-reduction alternatives, such as supervised diet, exercise and behavioral modification programs;
4. Be willing to commit to a long-term low calorie (1000-1500 calories/day) supervised diet;
5. Have reasonable weight loss expectations (accept a goal of losing up to 15% of body weight after 52 weeks);
6. Be able to follow requirements outlined in the protocol, including complying with the visit schedule and behavioral modification program, and willing to undergo protocol-specific procedures, e.g., endoscopy, local sedation, general anesthesia, upper gastrointestinal radiography (UGI), electrocardiography (EKG), gastric motility testing, and/or clinical laboratory testing, and must be willing to take prescribed proton pump inhibitors (PPIs);
7. Be able to provide written informed consent;
8. supporting that the subject is an appropriate study candidate;
9. Be willing to use contraception (e.g., birth control pills, condoms, abstinence) and avoid pregnancy during the study if female of child-bearing potential.

Exclusion Criteria:

1. Previous history of esophageal, gastric or duodenal surgery, any bariatric surgery, any hiatal hernia surgery, bowel obstruction surgery, adhesive peritonitis, and/or hiatal hernia > 4 cm;
2. A history of myocardial infarction in the previous 6 months: New York Heart Associate (NYHA) Class III or IV (heart failure) or cardiac arrhythmia (e.g. atrial fibrillation);
3. History or symptoms of varices, bowel obstruction, congenital or acquired GI anomalies (e.g., atresias, stenosis, stricture, and/or diverticula), severe renal, hepatic, and/or pulmonary disease;
4. History or symptoms of inflammatory bowel disease, such as Crohn's disease;
5. History of unstable thyroid disease;
6. History of uncontrolled gastro-esophageal reflux;
7. Type I diabetes;
8. History of dysphagia, esophageal stricture or esophageal food impaction;
9. Poor general health, in the opinion of the Placing and/or Evaluating Investigator, or presence of a specific medical condition that would increase the risks associated with endoscopy and/or placement of the device;
10. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
11. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD);
12. Specific diagnosed genetic or hormonal cause for obesity such as Prader Willi syndrome;
13. History or symptoms of esophageal or GI motility disorders (e.g., gastroparesis, achalasia, diffuse esophageal spasm) or symptoms of esophageal stricture;
14. Ongoing treatment with anticoagulants, steroids, aspirin > 100 mg, non-steroidal anti- inflammatory drugs (NSAIDS), or other medications known to be gastric irritants, and inability or unwillingness to discontinue the use of these concomitant medications;
15. Evidence of untreated psychiatric or eating disorders, such as major depression, schizophrenia, substance abuse;
16. Pregnancy, breast-feeding, or intention of becoming pregnant during the study (if female of childbearing potential);
17. A condition, or is in a situation, which in the Evaluating and/or Placing Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Percent change in total body weight (%TBL) . | 12 months
  Percent change in total body weight (%TBL) .

CONTACTS AND LOCATIONS:
Overall Officials: Evžen Machytka, MD, PhD, Principal Investigator — Asclepiades - Interna a Gastroenterologie, s.r.o.
Locations (1):
- Asclepiades - interna a gastroenterologie, s.r.o., Havířov, Czechia

IPD SHARING:
Plan to Share IPD: No
The authors have no plan make individual participant data available to other researchers